CLINICAL TRIAL: NCT05490472
Title: A Phase 1/2a, Multi-Center, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Evidence of Antitumor Activity of JAB-2485 in Adult Patients With Advanced Solid Tumors
Brief Title: JAB-2485 Activity in Adult Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jacobio Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JAB-2485-1001
Record Dates: First submitted 2022-07-25; First posted 2022-08-05 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumors; ER+ Breast Cancer; Triple Negative Breast Cancer, TNBC; ARID1A Gene Mutation; Small Cell Lung Cancer, SCLC
Keywords: Aurora A inhibitor; ARID1A Gene Mutation
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- JAB-2485 monotherapy, Phase 1, Dose Escalation (Experimental): Dose escalation of JAB-2485 will be administered as monotherapy to determine the MTD and RP2D.
  Interventions: Drug: JAB-2485 (Aurora A inhibitor)
- JAB-2485 monotherapy, Phase 2a, Dose Expansion (Experimental): JAB-2485 will be administered as monotherapy in patients with specific tumor types to evaluate the preliminary antitumor activity.
  Interventions: Drug: JAB-2485 (Aurora A inhibitor)

INTERVENTIONS:
Drug: JAB-2485 (Aurora A inhibitor) — Administered orally
  Arms: JAB-2485 monotherapy, Phase 1, Dose Escalation
Drug: JAB-2485 (Aurora A inhibitor) — Administered orally
  Arms: JAB-2485 monotherapy, Phase 2a, Dose Expansion

SUMMARY:
This study is to evaluate the safety and tolerability of JAB-2485 monotherapy in adult participants with advanced solid tumors.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of JAB-2485 monotherapy to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) during Dose Escalation phase when administered in participants with advanced solid tumors; then to further evaluate preliminary antitumor activity of JAB-2485 monotherapy at the RP2D during Dose Expansion phase in patients with advanced solid tumors such as ER+ breast cancer, triple negative breast cancer (TNBC), AT-rich interaction domain 1A (ARID1A) mutant solid tumors and small cell lung cancer (SCLC).

ELIGIBILITY:
Inclusion Criteria:

* Must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Must be able to provide an archived tumor sample
* Must have histologically or cytologically confirmed metastatic or locally advanced solid tumor

  * Dose Expansion phase cohorts must meet specific expression or gene mutation where indicated
* Must be refractory to or become intolerant of existing therapy(ies) known to provide clinical benefit for their condition
* Must have at least 1 measurable lesion per RECIST v1.1
* Must have adequate organ functions
* Must be able to swallow and retain orally administered medication

Exclusion Criteria:

* Has central nervous system (CNS) metastases or carcinomatous meningitis, except if CNS metastases treated and no evidence of radiographic progression or hemorrhage for at least 28 days
* Active infection requiring systemic treatment within 7 days
* Active hepatitis B virus (HBV), hepatitis C virus (HCV), or HIV
* Any severe and/or uncontrolled medical conditions
* left ventricular ejection fraction (LVEF) ≤50% assessed by echocardiogram (ECHO) or multigated acquisition scan (MUGA)
* QT interval using Fridericia's formula (QTcF) interval >470 msec
* Experiencing unresolved CTCAE 5.0 Grade >1 toxicities
* Clinically significant eye disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation phase: Number of participants with dose limiting toxicities (DLTs) | First 21 days of Cycle 1
  A DLT is defined as an adverse event (AE) regardless of attribution unless clearly related to underlying disease or extraneous cause during the first 21 days of Cycle 1 (DLT observation period).
Dose Escalation phase: Number of participants with adverse events (AEs) | Up to 3 years
  Participants will be assessed for incidence and severity of AEs according to NCI-CTCAE v5.0
Dose Expansion phase: Objective Response Rate (ORR) | Up to 3 years from baseline to RECIST confirmed Progressive Disease (PD)
  ORR is defined as the percentage of participants with partial response (PR) or complete response (CR) based on RECIST v1.1
Dose Expansion phase: Duration of Response (DOR) | Up to 3 years
  DOR is defined as the time from the participants initial objective response (CR or PR) to disease progression per CTCAE v1.1 or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Dose Escalation phase: Objective Response Rate (ORR) | Up to 3 years from baseline to RECIST confirmed Progressive Disease (PD)
  ORR is defined as the percentage of participants with PR or CR based on RECIST v1.1
Dose Escalation and Dose Expansion phase: Time to response (TTR) | Up to 3 years
  TTR is defined as the interval of time between the date of first treatment to the first documented response (CR or PR) as determined by investigator assessment per RECIST v1.1
Dose Escalation phase: Duration of Response (DOR) | Up to 3 years
  DOR is defined as the time from the participants initial objective response (CR or PR) to disease progression per CTCAE v1.1 or death due to any cause, whichever occurs first
Dose Escalation and Dose Expansion phase: peak plasma concentration (Cmax) | Up to 3 years
  Pharmacokinetic (PK) parameters of JAB-2485 monotherapy and the food effect assessment by using plasma or urine PK samples, including peak plasma concentration (Cmax)
Dose Escalation and Dose Expansion phase: time to peak plasma concentration(Tmax) | Up to 3 years
  Pharmacokinetic (PK) parameters of JAB-2485 monotherapy and the food effect assessment by using plasma or urine PK samples. Including time to peak plasma concentration (tmax)
Dose Escalation and Dose Expansion phase: Ctrough | Up to 3 years
  Pharmacokinetic (PK) parameters of JAB-2485 monotherapy and the food effect assessment by using plasma or urine PK samples. Including pre-dose through concentration (Ctrough)
Dose Escalation and Dose Expansion phase: Area under the curve (AUC) | Up to 3 years
  Pharmacokinetic (PK) parameters of JAB-2485 monotherapy and the food effect assessment by using plasma or urine PK samples. Including area under the plasma concentration versus time curve (AUC)
Dose Escalation and Dose Expansion phase: half-life (t½) | Up to 3 years
  Pharmacokinetic (PK) parameters of JAB-2485 monotherapy and the food effect assessment by using plasma or urine PK samples. Including half-life (t½)
Dose Escalation and Dose Expansion phase: total body clearance | Up to 3 years
  Pharmacokinetic (PK) parameters of JAB-2485 monotherapy and the food effect assessment by using plasma or urine PK samples. Including total body clearance
Dose Expansion phase: Progression Free Survival (PFS) | Up to 3 years
  PFS is defined as the interval of time between the date of first treatment to the earliest date of disease progression per RECIST v1.1 or death which occurs first.
Dose Expansion Phase 2a: Overall Survival (OS) | Up to 3 years
  OS is defined as the length of time between the date of first treatment to the date of death
Dose Expansion phase: Disease Control Rate (DCR) | Up to 3 years
  DCR is defined as percentage of participants with complete response (CR), partial response (PR), or stable disease (SD) per RECIST v1.1
Dose Expansion phase: Number of participants with adverse events (AEs) | Up to 3 years
  Participants will be assessed for incidence and severity of AEs according to NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (8):
- United States (4):
  - Henry Ford Health System, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Mary Crowley Cancer Research, Dallas, Texas
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
- China (4):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Jilin Cancer Hospital, Changchun, Jilin
  - Shandong Cancer Hospital, Jinan, Shandong